CLINICAL TRIAL: NCT07224997
Title: Trimethoprim-Sulfamethoxazole (TMP/SMX) Prophylaxis After Acute Kidney Injury to Prevent Post-discharge Infections
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Jonathan Samuel Chavez Iñiguez, Head of nephrology, Hospital Civil de Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Protocol CEI 214/25
Record Dates: First submitted 2025-10-27; First posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Acute Kidney Injuries; Acute Kidney Disease; Acute Kidney Injury (AKI)
MeSH Terms: conditions — Acute Kidney Injury | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Intervention Model Description: Experimental: TMP/SMX
  * Intervention: Drug: Trimethoprim-Sulfamethoxazole (TMP/SMX) 160/800 mg tablets every 48 hours
  * Dosing: One tablet by mouth, Trimethoprim-Sulfamethoxazole (TMP/SMX) 160/800 mg tablets every 48 hours, for 90 days post-discharge.
  * Other names: cotrimoxazole, sulfamethoxazole-trimethoprim. Bactrim F
  Placebo Comparator: Placebo
  * Intervention: Drug: Placebo (matching oral tablet)
  * Dosing: Matching schedule for 90 days post-discharge.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Arms & Interventions
  Experimental: TMP/SMX
  * Intervention: Drug: Trimethoprim-Sulfamethoxazole (TMP/SMX) 160/800 mg tablets every 48 hours
  * Dosing: One tablet by mouth, Trimethoprim-Sulfamethoxazole (TMP/SMX) 160/800 mg tablets every 48 hours, for 90 days post-discharge.
  * Other names: cotrimoxazole, sulfamethoxazole-trimethoprim. Bactrim F
  Placebo Comparator: Placebo
  * Intervention: Drug: Placebo (matching oral tablet)
  * Dosing: Matching schedule for 90 days post-discharge.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TMP/SMX (Experimental): Drug: Trimethoprim-Sulfamethoxazole (TMP/SMX) 160/800 mg tablets every 48 hours
  * Dosing: One tablet by mouth, Trimethoprim-Sulfamethoxazole (TMP/SMX) 160/800 mg tablets every 48 hours, for 90 days post-discharge.
  * Other names: cotrimoxazole, sulfamethoxazole-trimethoprim. Bactrim F
  Interventions: Drug: Drug: Trimethoprim-Sulfamethoxazole (TMP/SMX) 160/800 mg tablets every 48 hours
- Placebo (Placebo Comparator): Drug: Placebo (matching oral tablet)
  • Dosing: Matching schedule for 90 days post-discharge.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Drug: Trimethoprim-Sulfamethoxazole (TMP/SMX) 160/800 mg tablets every 48 hours — Drug: Trimethoprim-Sulfamethoxazole (TMP/SMX) 160/800 mg tablets every 48 hours
  • Dosing: One tablet by mouth, Trimethoprim-Sulfamethoxazole (TMP/SMX) 160/800 mg tablets every 48 hours, for 90 days post-discharge.
  Arms: TMP/SMX
Other: Placebo — Drug: Placebo (matching oral tablet)
  • Dosing: Matching schedule for 90 days post-discharge.
  Arms: Placebo

SUMMARY:
Official Title

Trimethoprim-Sulfamethoxazole (TMP/SMX) Prophylaxis After Acute Kidney Injury to Prevent Post-discharge Infections: A Randomized, Double-Blind, Placebo-Controlled Trial

Brief Summary

Acute kidney injury (AKI) is commonly followed by infections after hospital discharge. This randomized, double-blind, placebo-controlled trial will test whether prophylactic TMP/SMX reduces post-discharge infections in adults recently hospitalized with AKI. Participants will be randomized 1:1 to TMP/SMX or matching placebo and followed for 6 months. The primary outcome is the proportion of participants who develop any infection within 90 days after discharge. Secondary outcomes include time to first infection, infection-related hospitalization, mortality, safety/adverse events, and healthcare utilization through 180 days.

Detailed Description

Adults discharged after an index hospitalization complicated by AKI are at elevated infection risk. This trial evaluates whether short-term TMP/SMX prophylaxis reduces 90-day infections. After consent and eligibility confirmation near discharge, participants are randomized (1:1) to receive TMP/SMX or matching placebo with double-blind masking (participant and outcome assessor). Dosing is standardized per protocol. We will ascertain infections via structured follow-up, medical record review, and adjudication by blinded assessors. Safety monitoring will capture adverse events (e.g., rash, cytopenias, hyperkalemia). Analyses follow intention-to-treat.

Study Design

* Study Type: Interventional (Clinical Trial)
* Primary Purpose: Prevention
* Allocation: Randomized (1:1)
* Intervention Model: Parallel Assignment
* Masking: Double-blind (Participant, Outcomes Assessor)
* Estimated Enrollment: 60 patients per group
* Study Start Date: December 2025
* Primary Completion Date (Anticipated): January 2027 (last patient reaches 90-day outcome)
* Study Completion Date (Anticipated): July 2028 (last patient completes 180-day follow-up)

Arms & Interventions

Experimental: TMP/SMX

* Intervention: Drug: Trimethoprim-Sulfamethoxazole (TMP/SMX) 160/800 mg tablets every 48 hours
* Dosing: One tablet by mouth, Trimethoprim-Sulfamethoxazole (TMP/SMX) 160/800 mg tablets every 48 hours, for 90 days post-discharge.
* Other names: cotrimoxazole, sulfamethoxazole-trimethoprim. Bactrim F

Placebo Comparator: Placebo

* Intervention: Drug: Placebo (matching oral tablet)
* Dosing: Matching schedule for 90 days post-discharge.

Concomitant care: Allowed per treating clinician. Drug interactions and lab monitoring handled per protocol.

Outcome Measures

Primary Outcome

• Any infection within 90 days after discharge Time Frame: Day 0 (discharge) to Day 90 Measure: Proportion of participants with ≥1 infection, defined by clinical diagnosis requiring documentation (e.g., UTI, pneumonia, SSTI, bloodstream infection) and/or antimicrobial treatment initiation.

Secondary Outcomes

1. Time to first infection (days) within 90 days.
2. Infection-related hospitalization within 90 and 180 days.
3. All-cause mortality at 90 and 180 days.
4. Emergency department visits or unplanned readmissions within 180 days.
5. Antibiotic-related adverse events (rash, cytopenia, creatinine rise ≥0.3 mg/dL, hyperkalemia ≥5.5 mmol/L) through 180 days.
6. C. difficile infection within 180 days.
7. Recurrent AKI (KDIGO criteria) within 180 days.
8. Medication adherence (pill counts and/or self-report) over 90 days.
9. Major adverse kidney events over 90 days.

Eligibility Criteria

Inclusion Criteria

* Age ≥18 years.
* Index hospitalization complicated by AKI (KDIGO criteria) prior to discharge.
* Planned discharge to community/rehabilitation with capacity for follow-up.
* Ability to provide informed consent.

Exclusion Criteria

* Known allergy to sulfonamides or TMP/SMX.
* Pregnancy or breastfeeding.
* Severe hepatic disease (e.g., Child-Pugh C).
* Severe cytopenia (e.g., ANC <1.0×10⁹/L or platelets <50×10⁹/L).
* Baseline hyperkalemia (>5.5 mmol/L) not correctable prior to randomization.
* Concomitant medications with high-risk interactions not amenable to dose/monitoring (per protocol).
* Current systemic antimicrobial therapy planned for >14 days after discharge (prophylaxis not indicated).
* Inability to adhere to study procedures or follow-up.

Contacts/Locations

* Lead Sponsor / Responsible Party: Jonathan Samuel Chavez Iñiguez, Hospital Civil de Guadalajara, servicio de Nefrología
* Principal Investigator: Jonathan Samuel Chavez Iñiguez, Hospital Civil de Guadalajara, servicio de Nefrología, 3313299609
* Study Locations: Hospital Civil de Guadalajara, servicio de Nefrología, Hospital 278, colonia el Retiro. Guadalajara. Jalisco.

Ethics and Oversight

* Conducted in accordance with the Declaration of Helsinki and ICH-GCP.
* IRB/Ethics approval: Comité de etica en investigacion, Protocol CEI 214/25, Approval : October 16, 2025.
* Written informed consent obtained from all participants prior to any study procedures.
* Data

ELIGIBILITY:
Inclusion Criteria

* Age ≥18 years.
* Index hospitalization complicated by AKI (KDIGO criteria) prior to discharge.
* Planned discharge to community/rehabilitation with capacity for follow-up.
* Ability to provide informed consent.

Exclusion Criteria:

* Known allergy to sulfonamides or TMP/SMX.
* Pregnancy or breastfeeding.
* Severe hepatic disease (e.g., Child-Pugh C).
* Severe cytopenia (e.g., ANC <1.0×10⁹/L or platelets <50×10⁹/L).
* Baseline hyperkalemia (>5.5 mmol/L) not correctable prior to randomization.
* Concomitant medications with high-risk interactions not amenable to dose/monitoring (per protocol).
* Current systemic antimicrobial therapy planned for >14 days after discharge (prophylaxis not indicated).
* Inability to adhere to study procedures or follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Any infection within 90 days after discharge | Day 0 (discharge) to Day 90
  Proportion of participants with ≥1 infection, defined by clinical diagnosis requiring documentation (e.g., UTI, pneumonia, SSTI, bloodstream infection) and/or antimicrobial treatment initiation.

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data, protocol, SAP, and analytic code.
  * When: Within 12 months after primary results publication.
  * How: Upon reasonable request to the sponsor/PI and data-use agreement approval.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When: Within 12 months after primary results publication.
Access Criteria: How: Upon reasonable request to the sponsor/PI and data-use agreement approval.

DOCUMENTS (2):
  • Study Protocol (2025-11-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT07224997/Prot_000.pdf
  • Informed Consent Form (2025-11-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT07224997/ICF_001.pdf